CLINICAL TRIAL: NCT05958342
Title: CAlcium and VAsopressin Following Injury Early Resuscitation (CAVALIER) Trial
Acronym: CAVALIER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY23040043; W81XWH-6-D-0024 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Trauma; Hemorrhage
Keywords: hemorrhagic shock; trauma; calcium gluconate; vasopressin
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Shock, Hemorrhagic; Diabetes Insipidus | interventions — Calcium Gluconate; Vasopressins

STUDY DESIGN:
Intervention Model Description: In-Hospital phase: permuted block design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Prehospital Intervention Arm (Experimental): 1 gram calcium gluconate provided via intravenous or intraosseous access over approximately 2-5 minutes, initiated prior to trauma bay arrival and infused to completion following arrival if needed
  Interventions: Drug: Calcium Gluconate
- Prehospital Control Arm (Placebo Comparator): Identical volume saline placebo to prehospital intervention arm provided via intravenous or intraosseous access over approximately 2-5 minutes, initiated prior to trauma bay arrival and infused to completion following arrival if needed
  Interventions: Drug: saline placebo
- Early In-Hospital Intervention Arm (Experimental): 4-unit vasopressin bolus followed by a vasopressin infusion at 0.04 U/min for 8 hours. Administration of the bolus will be initiated as soon as feasible and within approximately 2 hours of enrollment. The infusion will be initiated within approximately 30 minutes of the bolus.
  Interventions: Drug: Vasopressin
- Early In-Hospital Control Arm (Placebo Comparator): volume matched saline bolus followed by volume matched normal saline placebo infusion for eight hours initiated within approximately two hours of enrollment
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: Calcium Gluconate — 1 gram calcium gluconate provided via intravenous or intraosseous access over approximately 2-5 minutes
  Arms: Prehospital Intervention Arm
Drug: Vasopressin — 4 unit vasopressin bolus followed by vasopressin infusion at 0.04 U/min for eight hours
  Arms: Early In-Hospital Intervention Arm
Drug: saline placebo — saline placebo volume matched to prehospital or in hospital phase
  Arms: Early In-Hospital Control Arm; Prehospital Control Arm

SUMMARY:
The CAlcium and VAsopressin following Injury Early Resuscitation (CAVALIER) Trial is a proposed 4 year, double-blind, mutli-center, prehospital and early in hospital phase randomized trial designed to determine the efficacy and safety of prehospital calcium and early in hospital vasopressin in patients at risk of hemorrhagic shock.

DETAILED DESCRIPTION:
Resuscitation strategies for the acutely injured patient in hemorrhagic shock have evolved. Patients benefit from receiving less crystalloid in favor of blood transfusions with balanced ratios of plasma and platelets or whole blood resuscitation. These resuscitation practices are termed Damage Control Resuscitation and have been incorporated into resuscitation protocols in Level I trauma centers across the country. Damage Control Resuscitation represents standard practice for military and civilian trauma. Despite these changes, deaths from traumatic hemorrhage continue to occur in the first hours following trauma center arrival, underscoring the importance of early, novel interventions.

Hypocalcemia following traumatic injury is exceedingly common following severe traumatic injury in patients at risk of hemorrhagic shock. During hemorrhagic shock resuscitation, pathways reliant upon calcium such as platelet function, intrinsic and extrinsic hemostasis, and cardiac contractility are disrupted. Citrate containing transfusion products are known to further reduce calcium levels through chelation during trauma resuscitation. Hypocalcemia has consistently been shown to be independently associated with the risk of large volume blood transfusion and mortality. Current management practices include calcium replacement during the in hospital phase of care in patients receiving blood products. Early calcium replacement in patients at risk of hemorrhage and hypocalcemia may mitigate coagulopathy, maintain hemostasis, improve hemodynamics and outcomes, and may reduce complications attributable to hemorrhagic shock.

Arginine vasopressin is a physiologic hormone released by the posterior pituitary in response to hypotension and is commonly used as a vasopressor for critically ill patients for the treatment of hypotension due to multiple causes including sepsis. Prolonged hemorrhagic shock has the potential to alter systemic vasomotor tone which can progress to refractory/recalcitrant hypotension. Patients receiving resuscitation for hemorrhage are at risk of vasopressin deficiency. Vasopressin may improve hemostasis by enhancing platelet function and augmenting clot formation. Vasopressin infusion soon after injury in patients in hemorrhagic shock has been demonstrated to be safe and result in a reduction in blood transfusion requirements and a lower incidence of deep venous thrombosis.

Whole blood, red cells, and blood components are a precious and limited resource. Trauma resuscitation adjuncts such as early calcium and vasopressin may provide benefit when transfusion products are limited and may provide additional benefit even when transfusion capabilities remain robust. Due to their action on coagulation and hemodynamic cascades in the injured patient, these resuscitation adjuncts have the potential to interact and provide additive benefit to the injured patient. However, safety and efficacy of prehospital calcium and early in hospital vasopressin remain inadequately characterized. Enrolled patients may participate in the prehospital phase (calcium), in-hospital phase (vasopressin), or both. The aims of the CAlcium and VAsopressin following Injury Early Resuscitation (CAVALIER) trial are to determine the efficacy and safety of prehospital calcium supplementation and early in hospital vasopressin infusion as compared to standard care resuscitation in patients at risk of hemorrhagic shock and to appropriately characterize any additive effect of both resuscitation adjunct interventions.

ELIGIBILITY:
Inclusion Criteria:

Prehospital Phase:

Injured patients at risk of hemorrhagic shock being transported from scene or referral hospital to a participating CAVALIER trial site who meet the following criteria:

1A. Systolic blood pressure ≤ 90mmHg and tachycardia (HR ≥ 108) at scene, at outside hospital, or during anticipated transport to a participating CAVALIER trial site

OR

1B. Systolic blood pressure ≤ 70mmHg at scene, at outside hospital, or during anticipated transport to a participating CAVALIER trial site

Early In-Hospital Phase:

Injured patients at a participating CAVALIER trial site at risk of hemorrhagic shock who meet the following criteria:

1A. Systolic blood pressure ≤ 90mmHg and tachycardia (HR ≥ 108) at scene, at outside hospital, during transport, or in emergency department of a participating CAVALIER trial site

OR

1B. Systolic blood pressure ≤ 70mmHg at scene, at outside hospital, during transport, or in emergency department of a participating CAVALIER trial site

AND

2.Blood/blood component transfusion initiated in prehospital setting or deemed clinically indicated within 60 minutes of arrival at the enrolling trauma center

AND 3. Clinical team deems Operating Room for major hemorrhage control procedure (e.g., laparotomy, thoracotomy, vascular exploration or extremity amputation) indicated within 60 minutes of arrival at the enrolling trauma center

AND

4. Anticipated admission to intensive care unit (ICU)

Exclusion Criteria:

Prehospital Phase

1. Wearing NO CAVALIER opt-out bracelet
2. Age > 90 or < 18 years of age
3. Isolated fall from standing injury mechanism
4. Known prisoner
5. Known pregnancy
6. Traumatic arrest with > 5 minutes of CPR without return of vital signs
7. Brain matter exposed or penetrating brain injury
8. Isolated drowning or hanging victims
9. Objection to study voiced by subject or family member at the scene or at the trauma center
10. Inability to obtain IV/IO access

Early In-Hospital Phase:

1. Wearing NO CAVALIER opt-out bracelet
2. Age > 90 or < 18 years of age
3. Isolated fall from standing injury mechanism
4. Known prisoner
5. Known pregnancy
6. Traumatic arrest with > 5 minutes of CPR without return of vital signs
7. Brain matter exposed or penetrating brain injury
8. Isolated drowning or hanging victims
9. Objection to study voiced by subject or family member at the scene or at the trauma center
10. Inability to obtain IV access

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 30-day mortality | from randomization to death or 30 days, whichever comes first
  all cause mortality within 30 days

SECONDARY OUTCOMES:
Number of participants with 6-hour mortality | from randomization to death or 6 hours, whichever comes first
  all cause mortality within 6 hours
Number of participants with 24-hour mortality | from randomization to death or 24 hours, whichever comes first
  all cause mortality within 24 hours
Number of participants with In-hospital mortality | In hospital mortality from time of randomization to death or 30 days, whichever comes first
  death prior to hospital discharge
Number of participants with Death from hemorrhage | from randomization to death or 30 days, whichever comes first
  Death from hemorrhage adjudicated by the site investigator
Number of participants with Death from brain injury | from randomization to death or 30 days, whichever comes first
  Death from brain injury adjudicated by the site investigator
Blood and blood component transfusion requirements in the initial 6 hours | from randomization to 6 hours
  number of units transfused and type
Blood and blood component transfusion requirements in the initial 24 hours | from randomization to 24 hours
  number of units transfused and type
Incidence of Multiple Organ Failure (MOF) | Scores determined daily until up to Day 7 or ICU discharge, whichever comes first
  Evaluated via the Denver Post injury Multiple Organ Failure Score, characterized as an incidence rate (percentage) and as MOF free days. Patients never admitted to ICU or with length of stay less than 48 hours will have a score of 0. A summary Denver score of >3 will be classified as MOF.
Incidence of nosocomial infection | from randomization to death or 30 days
  Utilizing the CDC criteria for diagnosis of hospital acquired pneumonia and blood stream infection
Time to hemostasis | hospital arrival to 4 hours
  Determined by ability to reach nadir transfusion requirement of 1 unit of red blood cells in a 60 minute period in the first 4 hours following arrival. In the absence of ability to obtain hemostasis within the first 4 hours, the patient will be designated "non-hemostasis"
Incidence of coagulopathy by thromboelastography (TEG) | within 4 hours of arrival plus or minus 12
  TEG date collected only when obtained as part of clinical
Incidence of coagulopathy by thromboelastography (TEG) | within 24 hours of arrival plus or minus 12
  TEG date collected only when obtained as part of clinical
ICU free days | From hospital arrival to death or 30 days
  number of days the patient is alive and not admitted to ICU subtracted from 30
Hospital free days | From hospital arrival to death or 30 days
  number of days the patient is alive and not admitted to hospital subtracted from 30
Ionized calcium measurements | Measured in the first 60 minutes (+/- 3 hours), when feasible, during early stage resuscitation in emergency department or operating room
  Ionized calcium collected as part of clinical care or as research lab

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Zuckerberg San Francisco General Hospital and Trauma Center at University of California, San Francisco, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - University of Miami, Miami, Florida
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Principal Investigator
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript
Access Criteria: Requests for data will be submitted in writing and reviewed by the Principal Investigator